CLINICAL TRIAL: NCT06754072
Title: Virtual Reality-Based Hand Rehabilitation for Post-Surgical Degenerative Cervical Myelopathy: A Pilot Study
Brief Title: Hand Dexterity Training in Degenerative Cervical Myelopathy (DCM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other); North Carolina State University (Other)
Responsible Party: Principal Investigator, Aditya Vedantam, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00044319; PI: Vedantam (Other Grant/Funding Number: Advancing a Healthier Wisconsin Endowment)
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Degenerative Cervical Myelopathy
Keywords: degenerative cervical myelopathy; virtual reality; hand dexterity; post-surgical rehabilitation; neurorehabilitation; cervical spine; eeg
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Training Group (Experimental): Participants completed virtual reality-based hand training using the virtual keyboard system.
  Interventions: Other: Virtual Keyboard (VK) System

INTERVENTIONS:
Other: Virtual Keyboard (VK) System — Participants underwent a 4-week training program comprising 12 one-hour sessions to enhance finger individuation and motor control using a virtual reality platform.

SUMMARY:
This clinical study aimed to evaluate the effectiveness of a virtual reality-based training intervention for improving hand dexterity and promoting neuroplasticity in individuals with Degenerative Cervical Myelopathy (DCM) after surgical decompression. Participants completed a 4-week training program using the Virtual Keyboard (VK) system, which facilitated repetitive, individualized finger movements in a virtual environment. Outcomes were measured pre- and post-training to quantify improvements in hand dexterity, quality of life, and cortical motor activity.

DETAILED DESCRIPTION:
Degenerative Cervical Myelopathy (DCM) is a leading cause of non-traumatic spinal cord injury, often resulting in impaired hand dexterity and diminished quality of life. Despite surgical decompression being the primary treatment, over 30% of individuals experience persistent functional disability due to a lack of targeted post-surgical rehabilitative interventions. This study sought to address this clinical gap by implementing and evaluating a virtual reality-based hand training intervention.

The central hypothesis was that an intensive, individualized training program using the Virtual Keyboard (VK) system would improve hand dexterity in individuals with DCM and that these functional gains would be supported by measurable changes in cortical motor activity.

Study Design

This single-arm interventional study recruited participants who had undergone cervical spine surgery within six months. A total of 25 participants were enrolled, each completing:

A 4-week training program consisting of 12 one-hour sessions using the VK system. The system provided engaging, interactive tasks designed to promote finger individuation and precise motor control through real-time visual and auditory feedback.

Pre- and post-training evaluations assessing functional, neurophysiological, and quality-of-life outcomes.

Specific Aims- Aim 1: Quantify improvements in hand dexterity after the training intervention. Hypothesis: Training with the VK system would significantly improve hand function as measured by the Jebsen-Taylor Hand Function Test (JTHFT) and other clinical metrics.

Approach: Baseline, post-training, and follow-up evaluations measured outcomes including JTHFT scores, pinch strength, and sensorimotor tests.

Aim 2: Assess neuroplastic changes associated with training. Hypothesis: The training program would enhance cortical motor activation and connectivity, reflected in changes in beta-band event-related desynchronization (ERD) and coherence measured via quantitative EEG (qEEG).

Approach: Participants underwent qEEG during finger-tapping tasks at each evaluation, and EEG data were analyzed for changes in cortical activation patterns.

Outcomes and Measures- Primary outcomes included: Improvement in hand function as measured by JTHFT scores and related clinical tests.

Changes in cortical motor activity and connectivity, including event-related desynchronization and coherence, derived from qEEG data.

Secondary outcomes included quality-of-life measures (SF-36 physical component score and EuroQol 5D).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Degenerative Cervical Myelopathy.
* Completed cervical spine surgery within 6 months.
* Modified Japanese Orthopaedic Association (mJOA) upper limb motor score between 1-4.

Exclusion Criteria:

* Pregnancy.
* History of brain or upper extremity surgery within the past year.
* Significant arm/hand pain limiting movement.
* Complete paralysis of the hands (mJOA=0).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Jebsen-Taylor Hand Function Test | Baseline, post-training and follow-up.
  The Jebsen-Taylor Hand Function Test (JTHFT) is a standardized test used to assess hand function during everyday activities. It consists of seven timed subtests, such as writing, card turning, and object manipulation. The outcome is recorded as the time taken to complete each task in seconds, where lower times indicate better hand function.

SECONDARY OUTCOMES:
Quantitative Electroencephalograms (qEEG) | Baseline, post-training and follow-up.
  Beta-band event-related desynchronization (ERD) and cortical coherence are key neural markers often analyzed during finger-tapping tasks to study motor control and cortical connectivity. These measures are often used in clinical studies (e.g., DCM, stroke) to evaluate motor system integrity and changes due to interventions or disease progression.
Nine-Hole Peg Test (9HPT) | Baseline, post-training and follow-up.
  The Nine-Hole Peg Test (9HPT) is a standardized test used to measure finger dexterity. It involves placing and removing pegs from nine holes as quickly as possible. The outcome is recorded as the time taken in seconds, where lower times indicate better dexterity.
Box and Blocks Test (BBT) | Baseline, post-training and follow-up.
  The Box and Blocks Test is a measure of gross manual dexterity. It involves moving as many blocks as possible from one compartment of a box to another in 60 seconds. The score is the total number of blocks moved, where higher scores indicate better manual dexterity.
QuickDASH | Baseline, post-training and follow-up.
  The QuickDASH is a subset of 11 items from the 30-item DASH (Disabilities of the Arm, Shoulder, and Hand) and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. Lower scores indicate better outcomes.
Three-point pinch strength | Baseline, post-training and follow-up.
  Sensorimotor hand function 3-point pinch strength using a pinch gauge (PG-60, B&L Engineering) measured in pounds (lbs.).
Touch sensitivity | Baseline, post-training (1 week after VK training), and 4-week follow-up ( 4 weeks after VK training).
  Touch sensitivity of the palmar and dorsal hand using von Frey filaments (Aesthesio®), scored out of 12 (12 indicates full sensation)
EuroQol 5-Dimension score | Baseline, post-training and follow-up.
  The EuroQol 5-Dimension (EQ-5D) is a standardized measure of health-related quality of life. The minimum level sum score (LSS) is derived by summing the responses across the five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each scored from 1 (no problems) to 3 (extreme problems) score is 5, and the maximum score is 15, where higher scores indicate worse health status. It also includes a Visual Analog Scale (VAS) scored from 0 to 100, where higher scores indicate better health.
Short Form-36 Health Survey version 2 | Baseline, post-training and follow-up.
  The Short Form-36 Health Survey version 2 (SF-36v2) is a validated, comprehensive measure of health-related quality of life. It includes eight domains (e.g., physical functioning-physical component score (PCS), and mental health-mental component score (MCS)) with scores ranging from 0 to 100, where higher scores indicate better health and functioning. An overall summary score for physical and mental health can also be derived.
Modified Japanese Orthopedic Association scale | Baseline, post-training and follow-up.
  The Modified Japanese Orthopaedic Association (mJOA) Score is a clinical scale used to evaluate the severity of cervical myelopathy. It assesses motor function in the upper and lower extremities, sensation, and bladder function. The total score ranges from 0 to 18, where higher scores indicate better neurological function and less severe disability.
Myelopathy Disability Index | Baseline, post-training and follow-up.
  The Myelopathy Disability Index (MDI) is a validated measure used to assess disability in individuals with cervical myelopathy. It consists of 10 items, each scored from 0 (no disability) to 10 (severe disability). The total score ranges from 0 to 100, where higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Vedantam, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Due to confidentiality and privacy concerns, individual participant data (IPD) will not be shared with other researchers. All study data will be presented in aggregate form in the final published results, with appropriate measures taken to ensure participant anonymity and data security.

REFERENCES:
- [Background] Thielbar KO, Lord TJ, Fischer HC, Lazzaro EC, Barth KC, Stoykov ME, Triandafilou KM, Kamper DG. Training finger individuation with a mechatronic-virtual reality system leads to improved fine motor control post-stroke. J Neuroeng Rehabil. 2014 Dec 26;11:171. doi: 10.1186/1743-0003-11-171. PMID 25542201

DOCUMENTS (1):
  • Informed Consent Form (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT06754072/ICF_000.pdf